CLINICAL TRIAL: NCT04000932
Title: Comparison of Local Steroid Injection With Platelet Rich Plasma in the Treatment of Carpal Tunnel Syndrome
Brief Title: Platelet Rich Plasma in Carpal Tunnel Syndrome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Sevgi Ikbali Afsar, Associate Professor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KA14/13
Record Dates: First submitted 2018-04-25; First posted 2019-06-27 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal tunnel syndrome; Injection; Platelet rich plasma
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Methods

STUDY DESIGN:
Intervention Model Description: prospective, randomized, controlled, double blind.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patient will not be informed about which group will be taken. Randomization will be performed by a simple randomization method by a researcher who is blind to the clinical and electrophysiological findings. The injection will be performed by a second researcher who is blind to the contents of the injection. The evaluations of the patients will be performed by a researcher who is blinded to the treatment applied and the initial assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet rich plasma (PRP) -T lab PRP kit (Experimental): A single 1ml PRP extract injection will be will be injected into the carpal tunnel of the wrist in which a diagnosis of carpel tunnel syndrome has been established. A 23 gauge needle will used to perform the injection through the distal wrist creased into the carpal tunnel. performed once into the carpal tunnel in the wrist . PRP will be obtained by centrifugation of autologous anticoagulated whole blood.
  Interventions: Drug: Local platelet rich plasma (PRP) injection-T-Lab PRP kit
- Diprospan ®, Schering Plough (Active Comparator): A single steroid injection (1 ml Diprospan ®, Schering Plough containing 6.43 mg of betamethasone dipropionate and 2.63 mg of betamethasone sodium phosphate) will be injected into the carpal tunnel of the wrist in which a diagnosis of carpel tunnel syndrome has been established. A 23 gauge needle will used to perform the injection through the distal wrist creased into the carpal tunnel.
  Interventions: Drug: Local steroid injection-Diprospan ®, Schering Plough

INTERVENTIONS:
Drug: Local platelet rich plasma (PRP) injection-T-Lab PRP kit — Platelet rich plasma (PRP) will be obtained by centrifugation of autologous anticoagulated whole blood. 1 ml PRP extract will be injected into the carpel tunnel (of the side with a diagnosis of carpel tunnel syndrome) via the distal wrist line using 23 gauge needle.
  Other Names: procedure
  Arms: Platelet rich plasma (PRP) -T lab PRP kit
Drug: Local steroid injection-Diprospan ®, Schering Plough — The local steroid injection ((1 ml Diprospan ®, Schering Plough containing 6.43 mg of betamethasone dipropionate and 2.63 mg of betamethasone sodium phosphate) will be performed once into the carpal tunnel.1 ml Diprospan ®, Schering Plough extract will be injected by using 23 gauge needle from the distal wrist line through the carpal tunnel only once.
  Other Names: procedure
  Arms: Diprospan ®, Schering Plough

SUMMARY:
The aim of this study is to evaluate the effect of local platelet rich plasma injection therapy in patients with mild to moderate idiopathic carpal tunnel syndrome (CTS) with clinical and electrophysiological parameters. Also the effect of platelet rich plasma and local steroid injection will be compared.

DETAILED DESCRIPTION:
Research sample; Voluntary female patients who are referred to the Physical Therapy and Rehabilitation Outpatient Clinic and who have a clinical and electrophysiological diagnosis of mild or moderate CTS. Patients aged between 25-70 years and who have complaints consistent with CTS for more than 3 months will be selected.

The size of the sample was determined by the preliminary statistical study conducted using the NCSS-PASS 12 program, and will consist of 84 patients.

Patients will be randomly allocated to one of two groups. Local platelet rich plasma (PRP) injection in the first group (n = 42) and local steroid injection in the second group (n = 42) will be performed once into the carpal tunnel. PRP will be obtained by centrifugation of autologous anticoagulated whole blood. 6.43 mg of betamethasone dipropionate and 2.63 mg of betamethasone sodium phosphate will be administered as local steroids. Both groups will be recommended a resting splint for use in the day time when possible and at night time. Clinical and electrophysiological evaluations of all patients will be performed by a researcher who is blinded to the treatment received by the patient. The electrophysiological and clinical evaluations of the patients will be done by the same investigator before and after the 1st and 3rd months of therapy. At one and three month follow up, Symptom severity and functional capacity will be assessed using the Boston Carpal Tunnel Syndrome Questionnaire. The hand grip strength of the patients will be assessed using a Jamar hand dynamometer ( (Baseline hydraulic hand dynomometer, Irvington, NY, USA) and the finger holding power by pinchmeter. Conventional motor and sensory nerve conduction studies will be applied as electrodiagnostic studies.

ELIGIBILITY:
Inclusion Criteria:

* female patient 25-75 years old
* Symptoms consistent with carpal tunnel syndrome for at least 3 months
* Clinical and electrophysiological diagnosis of mild to moderate carpal tunnel syndrome
* Written informed consent obtained

Exclusion Criteria:

* Electrophysiological diagnosis of proximal median nerve neuropathy, cervical radiculopathy, brachial plexopathy, thoracic outlet syndrome
* Those with a past medical history of diabetes mellitus, hypothyroidism, pregnancy, chronic inflammatory rheumatic disease, renal insufficiency which may predispose to CTS
* Patients with a history of wrist surgery or radius distal tip fracture
* Patients who underwent carpal tunnel local steroid injection within the previous 3 months
* Patients with a cardiac pacemaker
* History of hematological disease (coagulopathy) or patients receiving anticoagulant or antiaggregant therapy
* Severe cardiovascular disease
* Infection, immunosuppression
* Patients using non-steroidal anti-inflammatory drugs up to 5 days before PRP injection patients with hemoglobin levels below 11 and platelet levels below 150,000

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2018-07-15 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
median nerve sensory conduction velocity | 3 months
  median nerve sensory conduction velocity in the palm wrist segment

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Ikbali Afsar, Assoc Prof, Principal Investigator — Baskent University Faculty of Medicine
Locations (1):
- Baskent University Faculty of Medicine, Ankara Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mondelli M, Giannini F, Giacchi M. Carpal tunnel syndrome incidence in a general population. Neurology. 2002 Jan 22;58(2):289-94. doi: 10.1212/wnl.58.2.289. PMID 11805259
- [Background] Palmer KT, Harris EC, Coggon D. Carpal tunnel syndrome and its relation to occupation: a systematic literature review. Occup Med (Lond). 2007 Jan;57(1):57-66. doi: 10.1093/occmed/kql125. Epub 2006 Nov 2. PMID 17082517
- [Background] Piazzini DB, Aprile I, Ferrara PE, Bertolini C, Tonali P, Maggi L, Rabini A, Piantelli S, Padua L. A systematic review of conservative treatment of carpal tunnel syndrome. Clin Rehabil. 2007 Apr;21(4):299-314. doi: 10.1177/0269215507077294. PMID 17613571
- [Background] Özçete ZA, Öztürk C, Yağız OA, Hepgüler S, Atamaz FÇ. Kısa dalga tedavisinin idiopatik karpal tünel sendromundaki etkinliği: Randomize çift kör kontrollü çalışma. Türk Fiz Tıp Rehab Derg.2013;59:103-7.
- [Background] Park GY, Kwon DR. Platelet-rich plasma limits the nerve injury caused by 10% dextrose in the rabbit median nerve. Muscle Nerve. 2014 Jan;49(1):56-60. doi: 10.1002/mus.23863. Epub 2013 Sep 20. PMID 23558771
- [Background] Sariguney Y, Yavuzer R, Elmas C, Yenicesu I, Bolay H, Atabay K. Effect of platelet-rich plasma on peripheral nerve regeneration. J Reconstr Microsurg. 2008 Apr;24(3):159-67. doi: 10.1055/s-2008-1076752. Epub 2008 Apr 30. PMID 18452111
- [Background] Eppley BL, Woodell JE, Higgins J. Platelet quantification and growth factor analysis from platelet-rich plasma: implications for wound healing. Plast Reconstr Surg. 2004 Nov;114(6):1502-8. doi: 10.1097/01.prs.0000138251.07040.51. PMID 15509939
- [Background] Thanasas C, Papadimitriou G, Charalambidis C, Paraskevopoulos I, Papanikolaou A. Platelet-rich plasma versus autologous whole blood for the treatment of chronic lateral elbow epicondylitis: a randomized controlled clinical trial. Am J Sports Med. 2011 Oct;39(10):2130-4. doi: 10.1177/0363546511417113. Epub 2011 Aug 2. PMID 21813443
- [Background] Sanchez M, Yoshioka T, Ortega M, Delgado D, Anitua E. Ultrasound-guided platelet-rich plasma injections for the treatment of common peroneal nerve palsy associated with multiple ligament injuries of the knee. Knee Surg Sports Traumatol Arthrosc. 2014 May;22(5):1084-9. doi: 10.1007/s00167-013-2479-y. Epub 2013 Mar 22. PMID 23519544
- [Background] Emel E, Ergun SS, Kotan D, Gursoy EB, Parman Y, Zengin A, Nurten A. Effects of insulin-like growth factor-I and platelet-rich plasma on sciatic nerve crush injury in a rat model. J Neurosurg. 2011 Feb;114(2):522-8. doi: 10.3171/2010.9.JNS091928. Epub 2010 Oct 29. PMID 21029038
- [Background] Apel PJ, Ma J, Callahan M, Northam CN, Alton TB, Sonntag WE, Li Z. Effect of locally delivered IGF-1 on nerve regeneration during aging: an experimental study in rats. Muscle Nerve. 2010 Mar;41(3):335-41. doi: 10.1002/mus.21485. PMID 19802878
- [Background] Yu W, Wang J, Yin J. Platelet-rich plasma: a promising product for treatment of peripheral nerve regeneration after nerve injury. Int J Neurosci. 2011 Apr;121(4):176-80. doi: 10.3109/00207454.2010.544432. Epub 2011 Jan 19. PMID 21244302
- [Background] Jazayeri SM, Azizi S, Moghtaderi AR. Autologous blood injection in carpal tunnel syndrome (CTS). Electromyogr Clin Neurophysiol. 2009 Nov-Dec;49(8):369-72. PMID 20058545
- [Background] Stevens JC. AAEM minimonograph #26: the electrodiagnosis of carpal tunnel syndrome. American Association of Electrodiagnostic Medicine. Muscle Nerve. 1997 Dec;20(12):1477-86. doi: 10.1002/(sici)1097-4598(199712)20:123.0.co;2-5. PMID 9390659
- [Background] D'Arcy CA, McGee S. The rational clinical examination. Does this patient have carpal tunnel syndrome? JAMA. 2000 Jun 21;283(23):3110-7. doi: 10.1001/jama.283.23.3110. PMID 10865306
- [Derived] Senlikci HB, Afsar SI, Cosar SN, Kurtcebe AN, Ozen S, Yemisci OU. The effectiveness of single-dose blinded platelet-rich plasma (PRP) vs. corticosteroid injection in mild-to-moderate carpal tunnel syndrome: A prospective, randomized, double blind study. J Bodyw Mov Ther. 2025 Jun;42:995-1001. doi: 10.1016/j.jbmt.2025.01.057. Epub 2025 Jan 31. PMID 40325784